CLINICAL TRIAL: NCT06542744
Title: A Prospective, Multicentric, Randomized Clinical Investigation Assessing the Impact of Perineal Training With the Emagina Medical Device on Perineal Flexibility During Pregnancy and Childbirth
Brief Title: Comparison of the Flexibility of the Perineum in Primiparous Women Using the Medical Device Emagina During 90 Days of Their Pregnancy Compared to Those Having a Standard Pregnancy Follow-up
Acronym: PeriFlex
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mumming (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PeriFlex; 2023-A01980-45 (Other: Agence nationale de sécurité du médicament et des produits de santé)
Record Dates: First submitted 2024-07-30; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Pregnancy; Childbirth
Keywords: Pregnancy; Perineum; Perineal training; Perineal flexibility; Perineal trauma prevention; Pelvic floor disorder prevention; Delivery trauma; Episiotomies reduction; Perineal tearing prevention; Pelvic muscle injury; Vaginal delivery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects using the Emagina Medical device (Experimental): Emagina Medical device
  Interventions: Device: Training with the Emagina device at home until birth
- Control group (Other): Standard of Care (SOC)
  Interventions: Other: No intervention

INTERVENTIONS:
Device: Training with the Emagina device at home until birth — The subjects will use the device at home according to a series of 3 exercises, 2 sessions per week, followed by a series of 4 exercises, 3 sessions per week starting from D75.
  Arms: Subjects using the Emagina Medical device
Other: No intervention — The subjects will follow usual care instructions. Subjects are not trained in the use of Emagina.
  Arms: Control group

SUMMARY:
The goal of this clinical investigation is to learn if training with Emagina device can improve flexibility of the perineum during childbirth with the help of a balloon that inflates in the genital area according to a time-limited exercise program specifically developed to optimize results, in adult, pregnant women with their first child (single fetus) less than 24 weeks of amenorrhea at the time of inclusion (i.e. during the 5th month of pregnancy).

The main questions it aims to answer are:

* Does the Emagina training program improve perineal flexibility during pregnancy ?
* Does the Emagina training program reduce the proportion and importance of perineal tears, as well as the proportion of sutures and episiotomies during childbirth ?

Researchers will compare Emagina group to a Control group (no intervention) to see if Emagina device works to improve perineum flexibility.

Participants will :

* measure the flexibility of their perineum on 2 occasions 90 days apart, with or without perineal training
* perform perineal training with the Emagina medical device or follow current practice
* fill out e-questionnaires regarding quality of life, lifestyle, pelvic static disorders, sexual activity and urinary incontinence

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age
* Singleton (fetus)
* Primiparous subject
* Subject less than 5 months pregnant (between 20 and 24 week of amenorrhea)
* Subject affiliated to a social security plan
* Subject who has given written consent prior to any specific procedure related to the clinical investigation
* Subject able to understand and complete the clinical investigation questionnaires
* Subject having a smartphone and being able to download the Emagina app

Exclusion Criteria:

* High-risk pregnancy (subjects presenting pregnancy-related risks will be excluded from participating in this clinical investigation, including risks of premature delivery, cases of symptomatically low-lying placenta and any contraindications to sexual relations)
* Scheduled cesarean section prior to inclusion
* History of vaginal or perineal surgery prior to pregnancy
* Pelvic anomalies
* Threatened preterm delivery prior to inclusion
* Vaginismus
* Use of Epi-no prior to inclusion
* Collagenosis or other chronic disorders affecting collagen
* Planned home birth
* Nerve damage and other illnesses that reduce sensitivity to pain in the genital area (i.e. paraplegia, multiple sclerosis, diabetic neuropathy, medication that alters sensitivity in the genital area, vulvar varicose veins).
* Persons deprived of liberty, under guardianship or trusteeship
* Drug or alcohol abuse
* Dementia, mental impairment, or psychiatric pathology that may compromise subject informed consent and/or compliance with the protocol and trial monitoring
* Subject unable to comply with protocol monitoring for psychological, social, family or geographic reasons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Maximum diameter of balloon expelled at D90 | Day 90
  To compare the flexibility of the perineum in primiparous subject having followed, during the pregnancy, the program of perineal training of the medical device Emagina during 90 days versus those having had a standard pregnancy follow-up

SECONDARY OUTCOMES:
Comparison of the expulsive phase | At Birth
  Expulsive phase will be defined with: the duration of the expulsive phase, the % of instrumental extraction (forceps, spatulas or vacuum-assisted delivery), the % of epidural anesthesia
Comparison of perineal injuries | At birth
  Perineal injuries will be defined with: the degree of perineal tears (according to the classification of perineal trauma), the % of grades 1, 2, 3, 4, the % of episiotomies, the % of perineal suture
APGAR score of the baby at birth | At Birth
  APGAR score at 1 minute, 5 minutes and 10 minutes after birth
Height of the baby at birth | At birth
  Height measured in cm
Weight of the baby at birth | At birth
  Weight measured in g
Head size of the baby at birth | At birth
  Head circumference measured in cm
Sex of the baby | At birth
  Gender of the baby determined at birth
Quality of life (SF-12) | Baseline and 2 months after birth
  Quality of life assessed by the SF-12 and lifestyle assessed by a short survey
Subject's satisfaction during delivery | 2 months after birth
  Subject's satisfaction during delivery assessed by the QACE questionnaire
Postnatal pelvic statics disorders | At baseline and 2 months postpartum
  Pelvic statics disorders assessed by the PFIQ-7 questionnaire
Postnatal return to normal sexual activity | At baseline and 2 months postpartum
  The % of subjects with return to normal sexual activity 2 months after delivery assessed by FSFI questionnaire (Yes/No),
Postnatal urinary leakage | At baseline and 2 months postpartum
  the % of subjects with urinary leakage 2 months after delivery assessed by ICIQ-UI questionnaire
Postnatal perineal rehabilitation session | 2 months after birth
  Number of perineal rehabilitation session prescribed by investigator
Variation of pressure exerted by the perineum during the flexibility measurement | At Day 0 and Day 90 visits
  The variation of pressure exerted by the perineum during the flexibility measurement will be defined with following parameters: The pressure exerted while the balloon is fully inflated inside the vagina " IN ", The maximum pressure exerted during the expulsion of the balloon " EXP ", The pressure exerted when the balloon is outside " OUT ", Variation between IN and EXP defined as IN-EXP, Variation between EXP and OUT defined as EXP-OUT
Usability of the device | 2 months after birth
  Usability of Emagina assessed by the subjects through a questionnaire developed by the sponsor (i.e. ease of use of Emagina device, absence of technical issues while using Emagina device)
Percentage of Compliance with the device | From baseline to birth
  Percentage of Compliance assessed by the Emagina App and defined as the number of days of use divided on the theoretical days of use
Adverse events | From baseline through study completion, an average of 6 months
  Adverse events recorded from ICF (Informed Consent Form) signature until final visit including the rate of unscheduled cesarean sections

CONTACTS AND LOCATIONS:
Overall Officials: David Desseauve, MD, Principal Investigator — Centre Hospitalier Universitaire de Grenoble Alpes
Locations (15):
- France (15):
  - Ornella Ferrari, 1 Bis Rue Castéja, Boulogne-Billancourt
  - Annabelle Sallandre, 7 Rue Ambroise Paré, Coutances
  - Solène Baradu, 5 Rue des Sports, Grandchamps-des-Fontaines
  - Grazia Sabatino, 2 impasse du Gaz, Marseille
  - Jennifer Denys, 53 rue de la Méditerranée, Montpellier
  - Elsa Molinier, 127 Rue Maurice Béjart, Montpellier
  - Alexandra Sasportas, 8 Boulevard de Magenta, Paris
  - Alice Rault, 103 Avenue de la République, Paris
  - Marion Alglave, 8 Rue Ernest Renan, Paris
  - Sobiha Sbai, 370 Avenue Jean Jaurès, Ronchin
  - Tiphaine Cartier, 45 Boulevard des Belges, Rouen
  - Céline Vauclin, 1 Avenue Jacques Chastellain, Rouen
  - Ariane Gasulla, 43 Rue Camille Claudel, Saint-Paul-lès-Dax
  - Annabel Buzy, 39 avenue Jean Jaurès, Suresnes
  - Karen Methia, 15 Allée du Gros Chêne, Verneuil-sur-Seine